CLINICAL TRIAL: NCT04755829
Title: Breath Test to Predict Breast Cancer and Outcome of Mammography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Menssana Research, Inc. (Industry)
Collaborators: Mount Vernon Cancer Centre (Unknown); Zuyderland Medical Centre (Other); University of Erlangen-Nürnberg (Other)
Responsible Party: Sponsor
Other Study IDs: M2020 UK01
Record Dates: First submitted 2021-02-08; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer; Abnormal Mammogram, Unspecified
Keywords: screening mammography; biomarker of breast disease
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Normal screening mammogram (BIRADS 1 or 2)
  Interventions: Device: BreathX test for breath VOCs
- Group 2: Abnormal screening mammogram (BIRADS 3 to 6)
  Interventions: Device: BreathX test for breath VOCs

INTERVENTIONS:
Device: BreathX test for breath VOCs — Breath samples are collected into an ultra-clean bag and breath VOCs are analyzed with GC-SAW.

SUMMARY:
To validate a breath test that predicts risk of breast cancer and an abnormal mammogram.

DETAILED DESCRIPTION:
We will determine the accuracy of volatile organic compounds (VOCs) in the breath as predictors of risk of breast cancer and an abnormal mammogram. Breath samples will be collected using an ultra-clean collection bag and analyzed with gas chromatography surface acoustic wave detection (GC SAW)

The study will be performed in two phases:

Phase 1: Model-building phase (cross-sectional study): Breath VOCs will be employed to construct multivariate algorithms that distinguish between normal women and those with breast cancer and abnormal screening mammograms.

Phase 2: Model-testing phase (cross-sectional study): The predictive accuracy of these algorithms will be tested to predict outcomes in normal women and those with breast cancer and abnormal screening mammograms.

ELIGIBILITY:
Group 1: Normal screening mammogram

Inclusion Criteria:

1. Female aged 18 years or older
2. Understands the study, and is willing to give written informed consent to participate
3. If a screening mammogram was performed during the preceding six month period, then the results were reported as normal (BIRADS 1 or 2)
4. If a screening mammogram was not performed during the preceding six month period, then approves collection of the results of a screening mammogram if and when it is performed subsequently*.
5. Approves collection of relevant additional data for clinical research record if and when these data become available, including results of imaging studies, breast biopsy, and other relevant biomarker data e.g. status of BRCA1, BRCA2, HER2 and receptors (ER+ or ER-) and progesterone (PgR+ or PgR-) * If a subsequent screening mammogram is reported as abnormal, the subject will be transferred to Group 2 for analysis of data.

Exclusion Criteria:

1. Previous history of an abnormal mammogram, breast disease, or breast biopsy
2. Previous history of cancer of any site, with the exception of basal cell carcinoma of skin
3. Concurrent serious or potentially life-threatening disease (e.g. severe cardiac or infectious disease)
4. Concurrent acute pulmonary disease (e.g. influenza, influenza-like illness, acute asthma, or pneumonitis).
5. General anesthesia during the 10-day period prior to breath collection.

Group 2: Abnormal screening mammogram

Inclusion Criteria:

Female aged 18 years or older

1. Understands the study, and is willing to give written informed consent to participate
2. Abnormal screening mammogram during preceding six months (BIRADS 3-6)
3. Approves collection of relevant additional data for clinical research record if and when it becomes available, including results of imaging studies, biopsy results, and other relevant biomarker data e.g. status of BRCA1, BRCA2, HER2 and receptors (ER+ or ER-) and progesterone (PgR+ or PgR-)

Exclusion criteria:

1. Previous history of cancer of any site, with the exception of basal cell carcinoma of skin
2. Previous history of breast biopsy
3. Concurrent serious or potentially life-threatening disease (e.g. severe cardiac or infectious disease)
4. Concurrent acute pulmonary disease (e.g. influenza, influenza-like illness, acute asthma, or pneumonitis).
5. General anesthesia during the 10-day period prior to breath collection. -

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Phase 1 Model-building phase (unblinded)
  Subjects will be enrolled in two groups:
  Group 1. Normal screening mammogram (BIRADS 1 or 2) Group 2. Abnormal screening mammogram (BIRADS 3 to 6)
  Phase 2 Model-testing phase (blinded)
  Subjects will be enrolled in two groups:
  Group 3. Normal screening mammogram (BIRADS 1 or 2) Group 4. Abnormal screening mammogram (BIRADS 3 to 6)
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
BREATH TEST TO PREDICT BREAST CANCER | 2 years
  Determination of the sensitivity, specificity, and positive and negative predictive values of a breath test for biomarkers that predict the risk of an abnormal mammogram.
BREATH TEST TO PREDICT OUTCOME OF MAMMOGRAPHY | 2 years
  Determination of the sensitivity, specificity, and positive and negative predictive values of a breath test for biomarkers that predict the risk of an biopsy-proven breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Tenovici, Principal Investigator — Frimley Health NHS Foundation Trust; Marc Lobbes, MD, Principal Investigator — Zuyderland Medical Center; Peter Fasching, MD, Principal Investigator — University of Erlangen-Nürnberg
Locations (3):
- University of Erlangen, Erlangen, Germany
- Zuyderland Medical Center, Heerlen, Netherlands
- Frimley Health NHS Foundation Trust, Middlesex, United Kingdom

REFERENCES:
- [Background] Smith-Bindman R, Chu PW, Miglioretti DL, Sickles EA, Blanks R, Ballard-Barbash R, Bobo JK, Lee NC, Wallis MG, Patnick J, Kerlikowske K. Comparison of screening mammography in the United States and the United kingdom. JAMA. 2003 Oct 22;290(16):2129-37. doi: 10.1001/jama.290.16.2129. PMID 14570948
- [Background] Health, United States, 2015. Centers for Disease Control and Prevention National Center for Health Statistics; 2015.
- [Background] Jiang Y, Miglioretti DL, Metz CE, Schmidt RA. Breast cancer detection rate: designing imaging trials to demonstrate improvements. Radiology. 2007 May;243(2):360-7. doi: 10.1148/radiol.2432060253. PMID 17456866
- [Background] White A, Miller J, Royalty J, Ryerson AB, Benard V, Helsel W, Kammerer W. Clinical outcomes of mammography in the National Breast and Cervical Cancer Early Detection Program, 2009-2012. Cancer Causes Control. 2015 May;26(5):723-32. doi: 10.1007/s10552-015-0567-7. Epub 2015 Mar 26. PMID 25809209
- [Background] Welch HG, Passow HJ. Quantifying the benefits and harms of screening mammography. JAMA Intern Med. 2014 Mar;174(3):448-54. doi: 10.1001/jamainternmed.2013.13635. PMID 24380095
- [Background] Hackshaw A. Benefits and harms of mammography screening. BMJ. 2012 Jan 6;344:d8279. doi: 10.1136/bmj.d8279. No abstract available. PMID 22228697
- [Background] Kneepkens CM, Ferreira C, Lepage G, Roy CC. The hydrocarbon breath test in the study of lipid peroxidation: principles and practice. Clin Invest Med. 1992 Apr;15(2):163-86. PMID 1591898
- [Background] Kneepkens CM, Lepage G, Roy CC. The potential of the hydrocarbon breath test as a measure of lipid peroxidation. Free Radic Biol Med. 1994 Aug;17(2):127-60. doi: 10.1016/0891-5849(94)90110-4. PMID 7959173
- [Background] Aghdassi E, Allard JP. Breath alkanes as a marker of oxidative stress in different clinical conditions. Free Radic Biol Med. 2000 Mar 15;28(6):880-6. doi: 10.1016/s0891-5849(00)00189-1. PMID 10802218
- [Background] Spink DC, Katz BH, Hussain MM, Spink BC, Wu SJ, Liu N, Pause R, Kaminsky LS. Induction of CYP1A1 and CYP1B1 in T-47D human breast cancer cells by benzo[a]pyrene is diminished by arsenite. Drug Metab Dispos. 2002 Mar;30(3):262-9. doi: 10.1124/dmd.30.3.262. PMID 11854143
- [Background] Brueggemeier RW, Diaz-Cruz ES. Relationship between aromatase and cyclooxygenases in breast cancer: potential for new therapeutic approaches. Minerva Endocrinol. 2006 Mar;31(1):13-26. PMID 16498361
- [Background] Phillips M, Cataneo RN, Chaturvedi A, Kaplan PD, Libardoni M, Mundada M, Patel U, Zhang X. Detection of an extended human volatome with comprehensive two-dimensional gas chromatography time-of-flight mass spectrometry. PLoS One. 2013 Sep 25;8(9):e75274. doi: 10.1371/journal.pone.0075274. eCollection 2013. PMID 24086492
- [Background] Phillips M, Byrnes R, Cataneo RN, Chaturvedi A, Kaplan PD, Libardoni M, Mehta V, Mundada M, Patel U, Ramakrishna N, Schiff PB, Zhang X. Detection of volatile biomarkers of therapeutic radiation in breath. J Breath Res. 2013 Sep;7(3):036002. doi: 10.1088/1752-7155/7/3/036002. Epub 2013 Jun 24. PMID 23793046
- [Background] Qiao Y, Gao Z, Liu Y, Cheng Y, Yu M, Zhao L, Duan Y, Liu Y. Breath ketone testing: a new biomarker for diagnosis and therapeutic monitoring of diabetic ketosis. Biomed Res Int. 2014;2014:869186. doi: 10.1155/2014/869186. Epub 2014 May 11. PMID 24900994
- [Background] Amann A, Corradi M, Mazzone P, Mutti A. Lung cancer biomarkers in exhaled breath. Expert Rev Mol Diagn. 2011 Mar;11(2):207-17. doi: 10.1586/erm.10.112. PMID 21405971
- [Background] Phillips M, Altorki N, Austin JH, Cameron RB, Cataneo RN, Greenberg J, Kloss R, Maxfield RA, Munawar MI, Pass HI, Rashid A, Rom WN, Schmitt P. Prediction of lung cancer using volatile biomarkers in breath. Cancer Biomark. 2007;3(2):95-109. doi: 10.3233/cbm-2007-3204. PMID 17522431
- [Background] D'Amico A, Pennazza G, Santonico M, Martinelli E, Roscioni C, Galluccio G, Paolesse R, Di Natale C. An investigation on electronic nose diagnosis of lung cancer. Lung Cancer. 2010 May;68(2):170-6. doi: 10.1016/j.lungcan.2009.11.003. Epub 2009 Dec 2. PMID 19959252
- [Background] Montuschi P, Mores N, Trove A, Mondino C, Barnes PJ. The electronic nose in respiratory medicine. Respiration. 2013;85(1):72-84. doi: 10.1159/000340044. Epub 2012 Sep 25. PMID 23018197
- [Background] Ehmann R, Boedeker E, Friedrich U, Sagert J, Dippon J, Friedel G, Walles T. Canine scent detection in the diagnosis of lung cancer: revisiting a puzzling phenomenon. Eur Respir J. 2012 Mar;39(3):669-76. doi: 10.1183/09031936.00051711. Epub 2011 Aug 18. PMID 21852337
- [Background] Boedeker E, Friedel G, Walles T. Sniffer dogs as part of a bimodal bionic research approach to develop a lung cancer screening. Interact Cardiovasc Thorac Surg. 2012 May;14(5):511-5. doi: 10.1093/icvts/ivr070. Epub 2012 Feb 17. PMID 22345057
- [Background] Vijverberg SJ, Hilvering B, Raaijmakers JA, Lammers JW, Maitland-van der Zee AH, Koenderman L. Clinical utility of asthma biomarkers: from bench to bedside. Biologics. 2013;7:199-210. doi: 10.2147/BTT.S29976. Epub 2013 Aug 29. PMID 24009412
- [Background] Phillips M, Gleeson K, Hughes JM, Greenberg J, Cataneo RN, Baker L, McVay WP. Volatile organic compounds in breath as markers of lung cancer: a cross-sectional study. Lancet. 1999 Jun 5;353(9168):1930-3. doi: 10.1016/S0140-6736(98)07552-7. PMID 10371572
- [Background] Phillips M, Cataneo RN, Cummin AR, Gagliardi AJ, Gleeson K, Greenberg J, Maxfield RA, Rom WN. Detection of lung cancer with volatile markers in the breath. Chest. 2003 Jun;123(6):2115-23. doi: 10.1378/chest.123.6.2115. PMID 12796197
- [Background] Phillips M, Altorki N, Austin JH, Cameron RB, Cataneo RN, Kloss R, Maxfield RA, Munawar MI, Pass HI, Rashid A, Rom WN, Schmitt P, Wai J. Detection of lung cancer using weighted digital analysis of breath biomarkers. Clin Chim Acta. 2008 Jul 17;393(2):76-84. doi: 10.1016/j.cca.2008.02.021. Epub 2008 Mar 3. PMID 18420034
- [Background] Phillips M, Cataneo RN, Condos R, Ring Erickson GA, Greenberg J, La Bombardi V, Munawar MI, Tietje O. Volatile biomarkers of pulmonary tuberculosis in the breath. Tuberculosis (Edinb). 2007 Jan;87(1):44-52. doi: 10.1016/j.tube.2006.03.004. Epub 2006 Apr 25. PMID 16635588
- [Background] Phillips M, Basa-Dalay V, Bothamley G, Cataneo RN, Lam PK, Natividad MP, Schmitt P, Wai J. Breath biomarkers of active pulmonary tuberculosis. Tuberculosis (Edinb). 2010 Mar;90(2):145-51. doi: 10.1016/j.tube.2010.01.003. Epub 2010 Feb 26. PMID 20189456
- [Background] Phillips M, Boehmer JP, Cataneo RN, Cheema T, Eisen HJ, Fallon JT, Fisher PE, Gass A, Greenberg J, Kobashigawa J, Mancini D, Rayburn B, Zucker MJ. Prediction of heart transplant rejection with a breath test for markers of oxidative stress. Am J Cardiol. 2004 Dec 15;94(12):1593-4. doi: 10.1016/j.amjcard.2004.08.052. PMID 15589029
- [Background] Ludviksdottir D, Diamant Z, Alving K, Bjermer L, Malinovschi A. Clinical aspects of using exhaled NO in asthma diagnosis and management. Clin Respir J. 2012 Oct;6(4):193-207. doi: 10.1111/crj.12001. PMID 22898078
- [Background] Elitsur Y, Tolia V, Gilger MA, Reeves-Garcia J, Schmidt-Sommerfeld E, Opekun AR, El-Zimaity H, Graham DY, Enmei K. Urea breath test in children: the United States prospective, multicenter study. Helicobacter. 2009 Apr;14(2):134-40. doi: 10.1111/j.1523-5378.2009.00670.x. PMID 19298341
- [Background] Heartsbreath - H030004. 2004. at http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cftopic/pma/pma.cfm?num=H030004.
- [Background] Mathews JM, Raymer JH, Etheridge AS, Velez GR, Bucher JR. Do endogenous volatile organic chemicals measured in breath reflect and maintain CYP2E1 levels in vivo? Toxicol Appl Pharmacol. 1997 Oct;146(2):255-60. doi: 10.1006/taap.1997.8257. PMID 9344893
- [Background] Bulun SE, Lin Z, Zhao H, Lu M, Amin S, Reierstad S, Chen D. Regulation of aromatase expression in breast cancer tissue. Ann N Y Acad Sci. 2009 Feb;1155:121-31. doi: 10.1111/j.1749-6632.2009.03705.x. PMID 19250199
- [Background] Boots AW, van Berkel JJ, Dallinga JW, Smolinska A, Wouters EF, van Schooten FJ. The versatile use of exhaled volatile organic compounds in human health and disease. J Breath Res. 2012 Jun;6(2):027108. doi: 10.1088/1752-7155/6/2/027108. Epub 2012 May 23. PMID 22621865
- [Background] Phillips M, Beatty JD, Cataneo RN, Huston J, Kaplan PD, Lalisang RI, Lambin P, Lobbes MB, Mundada M, Pappas N, Patel U. Rapid point-of-care breath test for biomarkers of breast cancer and abnormal mammograms. PLoS One. 2014 Mar 5;9(3):e90226. doi: 10.1371/journal.pone.0090226. eCollection 2014. PMID 24599224
- [Background] Phillips M, inventor USPTO Application no. 20170188887. Ultra-clean bag or balloon for collection of volatile organic compounds in breath or air https://www.google.com/patents/US20170188887. USA2017.
- [Background] Phillips M. Method for the collection and assay of volatile organic compounds in breath. Anal Biochem. 1997 May 1;247(2):272-8. doi: 10.1006/abio.1997.2069. PMID 9177688
- [Background] Phillips M, Herrera J, Krishnan S, Zain M, Greenberg J, Cataneo RN. Variation in volatile organic compounds in the breath of normal humans. J Chromatogr B Biomed Sci Appl. 1999 Jun 11;729(1-2):75-88. doi: 10.1016/s0378-4347(99)00127-9. PMID 10410929